CLINICAL TRIAL: NCT01767207
Title: Mental Health and Cognitive Dysfunction: A Multicenter Study at Pediatric Rehabilitation Clinics in North Norway
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1009 (Rek)
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Patient Health Questionnaire; Mass Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- screening for mental disorders: screening for mental disorders
  Interventions: Other: mental disorders; Behavioral: screening for mental disorders

INTERVENTIONS:
Other: mental disorders — mental disorders
Behavioral: screening for mental disorders — screening for mental disorders

SUMMARY:
Patients referred to pediatric rehabilitation services have often cognitive deficits/intellectual disabilities.Neurocognitive assessment is, hence, important when designing treatment plans.

Children and adolescents with cognitive deficits and intellectual disabilities (ID) have a high risk of developing mental health problems. There is lack of knowledge about such comorbid mental disorders in the health service. There are also few validated instruments for assessing mental disorders among children and adolescents with cognitive deficits and ID both in Norway and abroad.

The main aims of the current multicentre study are to:

Investigate psychometric properties of different psychiatric instruments for children and adolescents. Investigate change and stability of symptoms over time. Investigate user satisfaction. The study will include Pediatric Rehabilitation Services at hospitals in Tromsø, Hammerfest and Bodø and will include in total 320 patients aged 4 to 18. We will use information from parents, teachers and patients, in addition to clinician-rated measures. Patients will be assessed at intake and after six months. We have conducted a pilot study in the period from 2012 to 2013.

DETAILED DESCRIPTION:
1. Investigate psychometric properties of a structured psychiatric interview

   (DAWBA) and a symptom measure (SDQ) in clinical samples of children and

   adolescents with cognitive deficits and intellectual disabilities. We will

   investigate the instruments' reliability and convergent validity with the

   Aberrant Behavior checklist (ABC), the DBC and the Social Responsiveness

   Scale (SRS), in addition to the clinician-rated severity of children's mental

   health problems measured with the CGAS and HoNOSCA.
2. The psychiatric instruments will be administrated at intake and after six

   months. We will investigate prevalence rates and indicators of disorder

   severity (comorbidity and persistence), including risk factors (socioeconomic

   status, parenting styles).
3. Investigate user satisfaction with the health service, i.e., the Pediatric

Rehabilitation Services.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 4 years to 18 years
2. Written informed consent to participate
3. Fluent in Norwegian
4. Normal or corrected to normal vision and hearing

   -

   Exclusion Criteria:

   -

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients referred to pediatric rehabilitation outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of mental disorders | Within the first or second day the patient is undergoing an assessment at the hospital
  The Development and Well Being Assessment (DAWBA) is a package of interviews, questionnaires and rating techniques designed to generate psychiatric diagnoses on 5-17 year old according to the International Statistical Classification of Diseases and Related Health Problems (ICD-10) and Diagnostic and Statistical Manual of Mental Disorders(DSM-IV).

SECONDARY OUTCOMES:
Prevalence of mental disorders | within 6 months after the initial assessment
  The Development and Well Being Assessment short-version is re-administered 6 months after taking part in the study (i.e., the basic outcome measure)

OTHER OUTCOMES:
Prevalence of maladaptive behavior | Within the first or second day the patient is undergoing an assessment at the hospital
  Aberrant Behavior Checklist
Current mental health status | Within the first or second day the patient is undergoing an assessment at the hospital
  Health of the Nation Outcome Scales for Children and Adolescents
General functioning of children | Within the first or second day the patient is undergoing an assessment at the hospital
  Children's Global Assessment
Prevalence of social impairment | Within the first or second day the patient is undergoing an assessment at the hospital
  Social Responsiveness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Halvorsen, PhD, Principal Investigator — University Hospital of North Norway
Locations (2):
- Norway (2):
  - Finnmarkssykehuset (The Finnmark Hospital Trust), Hammerfest
  - University Hospital of North Norway, Tromsø